CLINICAL TRIAL: NCT01155583
Title: A Phase I/II Trial Of Very Low to Low-Doses of Continuous Azacitidine in Combination With Standard Doses of Lenalidomide and Low-Dose Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Low-Dose Azacitidine, Lenalidomide, and Low-Dose Dexamethasone in Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE1A09; NCI-2010-01139 (Other: NCI/CTRP)
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-10

CONDITIONS: Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Azacitidine; Lenalidomide; Dexamethasone; Calcium Dobesilate; DNA Methylation; Gene Expression Profiling; Immunohistochemistry; Reverse Transcriptase Polymerase Chain Reaction; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - Azacitidine/Lenalidomide/Dexamethasone (Experimental): Dose Level (DL) 1 - Azacitidine 30mg/m2 1x week + Lenalidomide 25mg d1-21 every 28d + Dexamethasone 40mg once a week
  DL 2 - Azacitidine 40mg/m2 1x week + Lenalidomide 25mg d1-21 every 28d + Dexamethasone 40mg once a week
  DL 3 - Azacitidine 30mg/m2 2x week + Lenalidomide 25mg d1-21 every 28d + Dexamethasone 40mg once a week
  DL 4 - Azacitidine 40mg/m2 2x week + Lenalidomide 25mg d1-21 every 28d + Dexamethasone 40mg once a week
  DL 5 - Azacitidine 50mg/m2 2x week + Lenalidomide 25mg d1-21 every 28d + Dexamethasone 40mg once a week
  Patients (with GFR > 60 ml/min) receive azacitidine subcutaneously 1 or 2x per weekly and oral Dexamethasone 1x weekly starting on day 1. Patients receive oral lenalidomide 1x daily on days 1-21. Treatment repeats every 28 days for 6 courses. Patients then continue to receive lenalidomide as maintenance therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: azacitidine; Drug: lenalidomide; Drug: dexamethasone; Other: DNA methylation analysis; Other: gene expression analysis; Other: bone marrow aspiration; Other: immunohistochemistry staining method; Other: reverse transcriptase-polymerase chain reaction; Other: flow cytometry
- Arm B - Chronic Kidney Disease (CDK) Cohort (Experimental): DL (-1) - Azacitidine 30mg/m2 2x week + Lenalidomide 10mg d1-21 every 28d + Dexamethasone 40mg once a week
  DL 1 - Azacitidine 40mg/m2 2x week + Lenalidomide 10mg d1-21 every 28d + Dexamethasone 40mg once a week
  DL 2 - Azacitidine 50mg/m2 2x week + Lenalidomide 10mg d1-21 every 28d + Dexamethasone 40mg once a week
  Patients (with GFR 30-59 ml/min Chronic Kidney Disease (CKD)) receive azacitidine subcutaneously 1 or 2x per weekly and oral dexamethasone 1x weekly starting on day 1. Patients receive oral lenalidomide 1x daily on days 1-21. Treatment repeats every 28 days for 6 courses. Patients then continue to receive lenalidomide as maintenance therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: azacitidine; Drug: lenalidomide; Drug: dexamethasone; Other: DNA methylation analysis; Other: gene expression analysis; Other: bone marrow aspiration; Other: immunohistochemistry staining method; Other: reverse transcriptase-polymerase chain reaction; Other: flow cytometry

INTERVENTIONS:
Drug: azacitidine — Given by subcutaneous injection (SC)
  Other Names: 5-AC; 5-azacytidine; 5-AZC; azacytidine; ladakamycin; Vidaza
Drug: lenalidomide — Given orally
  Other Names: CC-5013; IMiD-1; Revlimid
Drug: dexamethasone — Given orally
  Other Names: Aeroseb-Dex; Decaderm; Decadron; Decaspray; DM; DXM
Other: DNA methylation analysis — Correlative studies
Other: gene expression analysis — Correlative studies
Other: bone marrow aspiration — Correlative studies
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Other: reverse transcriptase-polymerase chain reaction — Correlative studies
  Other Names: RT-PCR
Other: flow cytometry — Correlative studies

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as azacitidine and dexamethasone, work in different ways to stop the growth of cancer cells either by killing the cells or by stopping them from dividing. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Giving azacitidine together with lenalidomide and dexamethasone may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of azacitidine when given together with lenalidomide and low-dose dexamethasone in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Define the highest tolerated low dose (HTLD) and safety of azacitidine given at low but increasing doses up to 50mg/m2 twice a week concurrently with Glomerular filtration rate (GFR)-adjusted lenalidomide and low dose dexamethasone in patients with relapsed or refractory multiple myeloma.

SECONDARY OBJECTIVES:

* Response according to international response criteria (≥PR) and clinical benefit response (≥minor response according to adapted EBMT criteria)
* Correlate response with plasma activity of the azacitidine inactivating enzyme cytidine deaminase (CDA)
* Progression-free survival and overall survival
* Peripheral blood hematopoietic progenitor (CD34+) yield and time to neutrophil and platelet recovery in patients undergoing autologous stem cell transplantation
* Promoter demethylation and gene reactivation in myeloma cells and hematopoietic progenitors treated at the HTLD / HTLD-CKD level after cycle 1
* Changes in global gene expression in myeloma cells treated at the HTLD / HTLD-CKD level after cycle 1

OUTLINE:

This is a phase I, dose-escalation study of azacitidine followed by a phase II study.

Patients receive azacitidine subcutaneously once or twice weekly and oral dexamethasone once weekly starting on day 1. Patients also receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 6 courses. Patients then continue to receive lenalidomide as maintenance therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Refractory or relapsed multiple myeloma
* Measurable disease defined as at least one of the following: Serum m-spike ≥ 1g/dL, urine m-spike ≥ 200mg/24hrs, serum free light chains ≥ 100mg/L (provided the kappa/lambda ratio is abnormal), or bone marrow plasma cells ≥ 30%
* Previous therapy with IMiD™ compounds (thalidomide, lenalidomide, pomalidomide), proteasome inhibitors (bortezomib, carfilzomib), and corticosteroids must be discontinued at least 14 days before entry onto this study.
* Previous cytotoxic chemotherapy (e.g. alkylating chemotherapy, anthracyclines, and vinca alkaloids), radiation therapy to the pelvis, and any experimental therapy other than carfilzomib or pomalidomide must have been discontinued at least 28 days prior to entry onto this study.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2 at study entry.
* Laboratory test results within these ranges:

  * Absolute neutrophil count ≥ 1,500 /mm³
  * Platelet count ≥ 75,000/mm³
  * Calculated creatinine clearance (Cockcroft-Gault) ≥ 30ml/min.
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) levels ≤2 x ULN
* All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
* Females of childbearing potential (FCBP)must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin two acceptable methods of birth control, one highly effective method and one additional effective method at the same time, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin) if no additional risk factor for venous thromboembolic event (VTE) other than myeloma diagnosis according to IMW guidelines
* Able to take low molecular weight heparin or warfarin if ≥ 1 additional risk factor for VTE according to IMW guidelines

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Pregnant or breast feeding females (Lactating females must agree not to breast feed while taking lenalidomide or azacitidine)
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Use of any experimental drug or therapy other than carfilzomib and pomalidomide within 28 days of treatment start on this protocol.
* Neuropathy > Grade 2
* Known hypersensitivity to thalidomide, lenalidomide, azacitidine, or mannitol
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or lenalidomide drugs
* Concurrent use of other anti-cancer agents or treatments, concurrent radiation to the pelvis. Palliative radiation to areas outside the pelvis is allowed
* Previous inability to tolerate full-dose lenalidomide, adjusted to creatinine clearance (CrCl) according to Cockcroft-Gault at the time of previous lenalidomide treatment (25mg day 1-21 every 28 days if CrCl > 60ml/min, 10mg lenalidomide d1-21 every 28 days if CrCl < 60mL/min but > 30mL/min, lenalidomide 15mg every 48 h d1-21 every 28 days if CrCl < 30mL/min but not requiring dialysis, lenalidomide 5mg daily, day 1-21 every 28 days if CrCl < 30mL/min and requiring dialysis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-06; Primary Completion 2016-05-28 (Actual); Study Completion 2018-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Reu, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center; Ehsan Malek, MD, Principal Investigator — University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The 11 phase II participants were a separate population from phase I
Groups:
- Arm A (GFR>=60mL/Min) Dose Level DL 1: Azacitidine (AZA) 30mg/m2 1x week + Lenalidomide 25mg d1-21 every 28d + Dexamethasone 40mg once a week
  Azacitidine/Lenalidomide/Dexamethasone Patients receive azacitidine subcutaneously once or twice weekly and oral dexamethasone once weekly starting on day 1. Patients also receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 6 courses. Patients then continue to receive lenalidomide as maintenance therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
- Arm A (GFR>=60mL/Min) Dose Level 2: Azacitidine 40mg/m2 1x week + Lenalidomide 25mg d1-21 every 28d + Dexamethasone 40mg once a week Patients receive azacitidine subcutaneously once or twice weekly and oral dexamethasone once weekly starting on day 1. Patients also receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 6 courses. Patients then continue to receive lenalidomide as maintenance therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
- Arm A (GFR>=60mL/Min) Dose Level 3: Azacitidine 30mg/m2 2x week + Lenalidomide 25mg d1-21 every 28d + Dexamethasone 40mg once a week Patients receive azacitidine subcutaneously once or twice weekly and oral dexamethasone once weekly starting on day 1. Patients also receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 6 courses. Patients then continue to receive lenalidomide as maintenance therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
- Arm A (GFR>=60mL/Min) Dose Level 4: Azacitidine 40mg/m2 2x week + Lenalidomide 25mg d1-21 every 28d + Dexamethasone 40mg once a week Patients receive azacitidine subcutaneously once or twice weekly and oral dexamethasone once weekly starting on day 1. Patients also receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 6 courses. Patients then continue to receive lenalidomide as maintenance therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
- Arm A (GFR>=60mL/Min) Dose Level 5: Azacitidine 50mg/m2 2x week + Lenalidomide 25mg d1-21 every 28d + Dexamethasone 40mg once a week
  Patients receive azacitidine subcutaneously once or twice weekly and oral dexamethasone once weekly starting on day 1. Patients also receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 6 courses. Patients then continue to receive lenalidomide as maintenance therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
- Arm B (GFR 30-59mL/Min - CKD) Dose Level -1: Azacitidine 30mg/m2 2x week + Lenalidomide 10mg d1-21 every 28d + Dexamethasone 40mg once a week
  Patients receive azacitidine subcutaneously once or twice weekly and oral dexamethasone once weekly starting on day 1. Patients also receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 6 courses. Patients then continue to receive lenalidomide as maintenance therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
- Arm B (GFR 30-59mL/Min - CKD) Dose Level 1: Azacitidine 40mg/m2 2x week + Lenalidomide 10mg d1-21 every 28d + Dexamethasone 40mg once a week
- Arm B (GFR 30-59mL/Min - CKD) Dose Level 2: Azacitidine 50mg/m2 2x week + Lenalidomide 10mg d1-21 every 28d + Dexamethasone 40mg once a week
- Phase II Arm A or B GFR >= 30mL/Min Expansion Dose (50 BIW): Azacitidine 50mg/m2 2x week + Lenalidomide (10mg if CKD, 25mg if non-CKD) d1-21 every 28d + Dexamethasone 40mg once a week
Period: Phase I
Arm/Group | Arm A (GFR>=60mL/Min) Dose Level DL 1 | Arm A (GFR>=60mL/Min) Dose Level 2 | Arm A (GFR>=60mL/Min) Dose Level 3 | Arm A (GFR>=60mL/Min) Dose Level 4 | Arm A (GFR>=60mL/Min) Dose Level 5 | Arm B (GFR 30-59mL/Min - CKD) Dose Level -1 | Arm B (GFR 30-59mL/Min - CKD) Dose Level 1 | Arm B (GFR 30-59mL/Min - CKD) Dose Level 2 | Phase II Arm A or B GFR >= 30mL/Min Expansion Dose (50 BIW)
Started | 3 | 3 | 4 | 6 | 7 | 0 | 3 | 8 | 0
Completed | 3 | 3 | 4 | 6 | 6 | 0 | 3 | 5 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Not completed — Screen failure - did not start treatment | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Phase II - Expansion Phase
Arm/Group | Arm A (GFR>=60mL/Min) Dose Level DL 1 | Arm A (GFR>=60mL/Min) Dose Level 2 | Arm A (GFR>=60mL/Min) Dose Level 3 | Arm A (GFR>=60mL/Min) Dose Level 4 | Arm A (GFR>=60mL/Min) Dose Level 5 | Arm B (GFR 30-59mL/Min - CKD) Dose Level -1 | Arm B (GFR 30-59mL/Min - CKD) Dose Level 1 | Arm B (GFR 30-59mL/Min - CKD) Dose Level 2 | Phase II Arm A or B GFR >= 30mL/Min Expansion Dose (50 BIW)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who signed consent and were put on study
Groups:
- Arm A (GFR>=60mL/Min) Dose Level DL 1: Azacitidine (AZA) 30mg/m2 1x week + Lenalidomide 25mg d1-21 every 28d + Dexamethasone 40mg once a week Azacitidine/Lenalidomide/Dexamethasone Patients receive azacitidine subcutaneously once or twice weekly and oral dexamethasone once weekly starting on day 1. Patients also receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 6 courses. Patients then continue to receive lenalidomide as maintenance therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
  lenalidomide: Given orally
  dexamethasone: Given orally
  DNA methylation analysis: Correlative studies
  gene expression analysis: Correlative studies
  bone marrow aspiration: Correlative studies
  immunohistochemistry staining method: Correlative studies
  reverse transcriptase-polymerase chain reaction: Correlative studies
  flow cytometry: Correlative studies
- Arm A (GFR>=60mL/Min) Dose Level 2: Azacitidine 40mg/m2 1x week + Lenalidomide 25mg d1-21 every 28d + Dexamethasone 40mg once a week Patients receive azacitidine subcutaneously once or twice weekly and oral dexamethasone once weekly starting on day 1. Patients also receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 6 courses. Patients then continue to receive lenalidomide as maintenance therapy. Treatment continues in the absence of disease progression or unacceptable toxicity
  lenalidomide: Given orally
  dexamethasone: Given orally
  DNA methylation analysis: Correlative studies
  gene expression analysis: Correlative studies
  bone marrow aspiration: Correlative studies
  immunohistochemistry staining method: Correlative studies
  reverse transcriptase-polymerase chain reaction: Correlative studies
  flow cytometry: Correlative studies
- Arm A or B GFR >= 30mL/ Min Expansion Dose (50 BIW): Azacitidine 50mg/m2 2x week + Lenalidomide (10mg if CKD, 25mg if non-CKD) d1-21 every 28d + Dexamethasone 40mg once a week
- Total: Total of all reporting groups
Arm/Group | Arm A (GFR>=60mL/Min) Dose Level DL 1 | Arm A (GFR>=60mL/Min) Dose Level 2 | Arm A (GFR>=60mL/Min) Dose Level 3 | Arm A (GFR>=60mL/Min) Dose Level 4 | Arm A (GFR>=60mL/Min) Dose Level 5 | Arm B (GFR 30-59mL/Min - CKD) Dose Level -1 | Arm B (GFR 30-59mL/Min - CKD) Dose Level 1 | Arm B (GFR 30-59mL/Min - CKD) Dose Level 2 | Arm A or B GFR >= 30mL/ Min Expansion Dose (50 BIW) | Total
Number analyzed (Participants) | 3 | 3 | 4 | 6 | 7 | 0 | 3 | 7 | 11 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 2 | 4 | 4 | 0 | 0 | 3 | 6 | 23
  >=65 years | 1 | 1 | 2 | 2 | 3 | 0 | 3 | 4 | 5 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 2 | 4 | 0 | 1 | 5 | 8 | 25
  Male | 2 | 1 | 2 | 4 | 3 | 0 | 2 | 2 | 3 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 0 | 2 | 6 | 7 | 0 | 3 | 7 | 11 | 39
  Unknown or Not Reported | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 4
  White | 3 | 3 | 3 | 6 | 5 | 0 | 3 | 6 | 11 | 40
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 6 | 7 |  | 3 | 7 | 11 | 44

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Highest Tolerated Low Dose (HTLD)
Description: Azacitidine given at low but increasing doses up to 50mg/m2 twice a week. Maximum tolerated dose reported.
Time Frame: During the first 28-day cycle
Population: Participants in phase 1 portion of study
Measure: Number; unit: mg/m^2
Groups:
- Arm A - Azacitidine/Lenalidomide/Dexamethasone; Arm B - CKD Azacitidine/Lenalidomide/Dexamethasone: Patients receive azacitidine subcutaneously once or twice weekly and oral dexamethasone once weekly starting on day 1. Patients also receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 6 courses. Patients then continue to receive lenalidomide as maintenance therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
  azacitidine: Given SC
  lenalidomide: Given orally
  dexamethasone: Given orally
  DNA methylation analysis: Correlative studies
  gene expression analysis: Correlative studies
  bone marrow aspiration: Correlative studies
  immunohistochemistry staining method: Correlative studies
  reverse transcriptase-polymerase chain reaction: Correlative studies
  flow cytometry: Correlative studies
Arm/Group | Arm A - Azacitidine/Lenalidomide/Dexamethasone | Arm B - CKD Azacitidine/Lenalidomide/Dexamethasone
Number analyzed (Participants) | 23 | 11
mg/m^2 | 50 | 50

2. Secondary Outcome: Percent of Participants With Clinical Benefit and Response According to International Response Criteria
Description: Percent of participants with response according to international response criteria (>= PR) and percent of participants with clinical benefit response (>= minor response according to adapted EBMT criteria). Determined with serum and 24 hour urine protein electrophoresis, and as appropriate, supplemented by immunofixation, serum free light chain assay, and bone marrow examination. Response before high dose melphalan and autologous stem cell transplant will also be confirmed by two separate blood and 24 hour urine tests between the last dose of combination therapy and the first dose of the mobilizing agent.
Time Frame: at 6 months
Population: Response-evaluable participants. Data from different dose levels were combined for the analysis as pre-specified in the study protocol
Measure: Number; unit: percentage of participants
Groups:
- Overall Study - (Azacitidine/Lenalidomide/Dexamethasone): Participants receive azacitidine subcutaneously once or twice weekly and oral dexamethasone once weekly starting on day 1. Participants also receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 6 courses. Participants then continue to receive lenalidomide as maintenance therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
- Participants Who Received HTLD/HTLD-CKD: Participants treated with the HTLD and HTLD-CKD dose: Azacitidine 50mg/m2 2x week + Lenalidomide 25mg (or 10mg for CKD) d1-21 every 28d + Dexamethasone 40mg once a week
Arm/Group | Overall Study - (Azacitidine/Lenalidomide/Dexamethasone) | Participants Who Received HTLD/HTLD-CKD
Number analyzed (Participants) | 41 | 22
percentage of participants
  international response criteria (>= PR) | 20 | 23
  clinical benefit response (>= minor response) | 32 | 32

3. Secondary Outcome: Percent of Participants With Clinical Benefit and Response According to International Response Criteria
Description: as for outcome 2
Time Frame: at 12 months
Population: Response-evaluable participants
Measure: Number; unit: percentage of participants
Groups:
- Participants Who Received HTLD/HTLD-CKD: Participants who received HTLD and HTLD-CKD dose: Azacitidine 50mg/m2 2x week + Lenalidomide 25mg (or 10mg for CKD) d1-21 every 28d + Dexamethasone 40mg once a week
Arm/Group | Overall Study - (Azacitidine/Lenalidomide/Dexamethasone) | Participants Who Received HTLD/HTLD-CKD
Number analyzed (Participants) | 41 | 22
percentage of participants
  International response criteria (>= PR) | 22 | 23
  clinical benefit response (>= minor response) | 32 | 32

4. Secondary Outcome: Median Progression-free Survival (PFS)
Description: Median PFS, measured in months from study entry to progression as defined by international response criteria or death of any cause, whichever comes first
Time Frame: Up to 3 years
Population: Evaluable participants who received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Overall Study - (Azacitidine/Lenalidomide/Dexamethasone)
Number analyzed (Participants) | 42
months | 3.1 [2.1 to 5.1]

5. Secondary Outcome: Overall Survival
Description: Overall survival will be measured from study entry to death from any cause - median months survival will be reported
Time Frame: up to 3 years
Population: Evaluable participants who received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Overall Study - (Azacitidine/Lenalidomide/Dexamethasone)
Number analyzed (Participants) | 42
months | 18.6 [9.5 to 23.4]

6. Other Pre Specified Outcome: Changes in Global Gene Expression
Description: The RNA harvested from myeloma cells before and after the first cycle of therapy at the HTLD level will furthermore be used to identify changes in global gene expression using the Illumina® HT12 array.
Time Frame: before and after the first cycle of therapy
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Quantify the Activity of Azacitidine Inactivating Enzyme Cytidine Deaminase (CDA)
Description: Plasma from peripheral blood draws will be used to quantify the activity of CDA using an HPLC method.The enzymatic activity is determined by comparison of cytidine deamination achieved by plasma samples with deamination achieved by incubation of cytidine with dilutions of pure CDA enzyme standards.
Time Frame: at 6 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Promoter Demethylation and Gene Reactivation
Description: Promoter demethylation and gene reactivation will be measured at least at the HTLD level using the Illumina® HumanMethylation27 BeadChip array on CD138 purified and CD34 purified cells obtained from bone marrow aspirates
Time Frame: within 7 days before treatment start and at the end of cycle #1
Reporting Status: Not Posted

9. Other Pre Specified Outcome: CD34+ Cell Yield and Time to Neutrophil and Platelet Recovery
Description: CD34+ cell yield will be calculated based on flow cytometry of mononuclear cells harvested following stem cell mobilization. Time to neutrophil (> 1,000/mm3) and platelet (> 100,000/mm3) recovery will be counted from the day of stem cell infusion (=day 0)
Time Frame: after cycle 1 (28 days)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 3 years from study entry
Description: Participants who started treatment on study were followed for Adverse Events. Number of participants at risk on Arm B Dose Level -1 is 0 because no participants were accrued to this dose level.
Groups:
- Arm A (GFR>=60mL/ Min) Dose Level 2: Azacitidine 40mg/m2 1x week + Lenalidomide 25mg d1-21 every 28d + Dexamethasone 40mg once a week Patients receive azacitidine subcutaneously once or twice weekly and oral dexamethasone once weekly starting on day 1. Patients also receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 6 courses. Patients then continue to receive lenalidomide as maintenance therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
- Arm A (GFR>=60mL/ Min) Dose Level 3: Azacitidine 30mg/m2 2x week + Lenalidomide 25mg d1-21 every 28d + Dexamethasone 40mg once a week Patients receive azacitidine subcutaneously once or twice weekly and oral dexamethasone once weekly starting on day 1. Patients also receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 6 courses. Patients then continue to receive lenalidomide as maintenance therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
- Arm A (GFR>=60mL/ Min) Dose Level 4: Azacitidine 40mg/m2 2x week + Lenalidomide 25mg d1-21 every 28d + Dexamethasone 40mg once a week Patients receive azacitidine subcutaneously once or twice weekly and oral dexamethasone once weekly starting on day 1. Patients also receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 6 courses. Patients then continue to receive lenalidomide as maintenance therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
- Arm A (GFR>=60mL/ Min) Dose Level 5: Azacitidine 50mg/m2 2x week + Lenalidomide 25mg d1-21 every 28d + Dexamethasone 40mg once a week
  Patients receive azacitidine subcutaneously once or twice weekly and oral dexamethasone once weekly starting on day 1. Patients also receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 6 courses. Patients then continue to receive lenalidomide as maintenance therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm A (GFR>=60mL/Min) Dose Level DL 1 | Arm A (GFR>=60mL/ Min) Dose Level 2 | Arm A (GFR>=60mL/ Min) Dose Level 3 | Arm A (GFR>=60mL/ Min) Dose Level 4 | Arm A (GFR>=60mL/ Min) Dose Level 5 | Arm B (GFR 30-59mL/Min - CKD) Dose Level -1 | Arm B (GFR 30-59mL/Min - CKD) Dose Level 1 | Arm B (GFR 30-59mL/Min - CKD) Dose Level 2 | Arm A or B GFR >= 30mL/ Min Expansion Dose (50 BIW)
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 5/6 | 6/6 | 0/0 | 3/3 | 5/6 | 10/11
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 2/4 | 2/6 | 1/6 | 0/0 | 1/3 | 1/6 | 1/11
Other Adverse Events (participants affected / at risk) | 3/3 | 1/3 | 2/4 | 2/6 | 3/6 | 0/0 | 1/3 | 4/6 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (GFR>=60mL/Min) Dose Level DL 1 (N=3) | Arm A (GFR>=60mL/ Min) Dose Level 2 (N=3) | Arm A (GFR>=60mL/ Min) Dose Level 3 (N=4) | Arm A (GFR>=60mL/ Min) Dose Level 4 (N=6) | Arm A (GFR>=60mL/ Min) Dose Level 5 (N=6) | Arm B (GFR 30-59mL/Min - CKD) Dose Level -1 (N=0) | Arm B (GFR 30-59mL/Min - CKD) Dose Level 1 (N=3) | Arm B (GFR 30-59mL/Min - CKD) Dose Level 2 (N=6) | Arm A or B GFR >= 30mL/ Min Expansion Dose (50 BIW) (N=11)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (GFR>=60mL/Min) Dose Level DL 1 (N=3) | Arm A (GFR>=60mL/ Min) Dose Level 2 (N=3) | Arm A (GFR>=60mL/ Min) Dose Level 3 (N=4) | Arm A (GFR>=60mL/ Min) Dose Level 4 (N=6) | Arm A (GFR>=60mL/ Min) Dose Level 5 (N=6) | Arm B (GFR 30-59mL/Min - CKD) Dose Level -1 (N=0) | Arm B (GFR 30-59mL/Min - CKD) Dose Level 1 (N=3) | Arm B (GFR 30-59mL/Min - CKD) Dose Level 2 (N=6) | Arm A or B GFR >= 30mL/ Min Expansion Dose (50 BIW) (N=11)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (4) | 0 (0) | 0 (0) | 3 (17) | 3 (21)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 2 (4)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (12) | 2 (13)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (6)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (13) | 2 (28)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (6) | 2 (8) | 2 (15) | 0 (0) | 1 (1) | 4 (13) | 9 (29)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (4) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (30)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (22) | 2 (20)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (9) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 1 (5)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (10) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Itching scalp (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-07-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT01155583/Prot_SAP_000.pdf
  • Informed Consent Form (2016-02-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT01155583/ICF_001.pdf